CLINICAL TRIAL: NCT00814619
Title: Neoadjuvant Radiotherapy and Capecitabine With or Without Panitumumab in Patients With Advanced, K-ras Unmutated Rectal Cancer. A Randomized Multicenter Phase II Trial
Brief Title: Capecitabine and Radiation Therapy With or Without Panitumumab in Treating Patients With Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/07; SWS-SAKK-41-07; EudraCT-2008-006012-38; EU-20894; CDR0000629101
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage III rectal cancer; stage II rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Capecitabine; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive panitumumab IV over 30-90 minutes on days 1, 15, 29, 43, and 57 and oral capecitabine twice daily on days 8-40. Beginning on day 8, patients undergo daily fractions of 3-D conformal radiotherapy 5 days a week for 5 weeks. Beginning approximately 6 weeks after completion of panitumumab and chemoradiotherapy, patients undergo surgery.
  Interventions: Biological: panitumumab; Drug: capecitabine; Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy
- Arm II (Active Comparator): Patients receive oral capecitabine twice daily on days 1-33. Patients undergo concurrent 3-D conformal radiotherapy 5 days a week for 5 weeks. Beginning 6 weeks after completion of chemoradiotherapy, patients undergo surgery.
  Interventions: Drug: capecitabine; Procedure: therapeutic conventional surgery; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Biological: panitumumab — Given IV
  Other Names: Vectibix
  Arms: Arm I
Drug: capecitabine — Given orally
  Other Names: Xeloda
Procedure: therapeutic conventional surgery — Patients undergo surgical resection
Radiation: 3-dimensional conformal radiation therapy — Patients undergo radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy that uses a 3-dimensional (3-D) image of the tumor to help focus thin beams of radiation directly on the tumor, and giving radiation therapy in higher doses over a shorter period of time, may kill more tumor cells and have fewer side effects. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving capecitabine together with 3-D conformal radiation therapy is more effective with or without panitumumab in treating patients with advanced rectal cancer.

PURPOSE: This randomized phase II trial is studying giving capecitabine together with radiation therapy to see how well it works with or without panitumumab in treating patients with advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the efficacy and safety of neoadjuvant capecitabine and concurrent 3-dimensional conformal radiotherapy with vs without panitumumab in patients with advanced K-ras unmutated rectal cancer.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, T stage (T3 vs T4), tumor localization measured from caudal part of the tumor to the anocutaneous line (< 10 cm vs ≥ 10 cm), and number of EGFR gene copies (< 2.9 vs ≥ 2.9). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive panitumumab IV over 30-90 minutes on days 1, 15, 29, 43, and 57 and oral capecitabine twice daily on days 8-40. Beginning on day 8, patients undergo daily fractions of 3-D conformal radiotherapy 5 days a week for 5 weeks. Beginning approximately 6 weeks after completion of panitumumab and chemoradiotherapy, patients undergo surgery.
* Arm II: Patients receive oral capecitabine twice daily on days 1-33. Patients undergo concurrent 3-D conformal radiotherapy 5 days a week for 5 weeks. Beginning 6 weeks after completion of chemoradiotherapy, patients undergo surgery.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced adenocarcinoma of the rectum with or without nodal involvement

  * Stage mrT3-4 and/or mrN1-2, M0
  * Tumors must express wild type K-ras gene
* No distant metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Able to undergo surgery
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 100 g/L
* Creatinine clearance ≥ 50 mL/min
* AST ≤ 2.5 times upper limit normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must agree to use effective contraception during and for 12 months after completion of study
* No malignancy within the past 5 years with the exception of adequately treated cervical carcinoma in situ or localized nonmelanoma skin cancer
* No psychiatric disorder that would preclude understanding study-related information, giving informed consent, or complying with oral drug intake
* No prior existing conditions that would preclude radiotherapy
* No clinically significant (i.e., active) cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, and cardiac arrhythmia even if controlled with medication) or myocardial infarction within the past 12 months
* No lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* No serious underlying medical condition that, in the judgement of the investigator, could impair the ability of the patient to participate in the trial (e.g., active autoimmune disease or uncontrolled diabetes)
* No known dihydropyrimidine dehydrogenase deficiency
* No known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior treatment in a clinical trial
* No other concurrent experimental drugs, anticancer therapy, or investigational treatments
* No prior treatment for rectal cancer
* No prior anti-EGFR antibody therapy (e.g., cetuximab) or small-molecule EGFR inhibitors (e.g., erlotinib hydrochloride)
* No concurrent treatment with brivudine, lamivudine, ribavirin, or any other nucleoside analogues
* No organ allografts
* No concurrent drugs contraindicated for use with the trial drugs
* No other concurrent anti-EGFR-targeting agents
* No other concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pathological complete or near-complete response (Dworak grade 3 and 4) | after 13 weeks.

SECONDARY OUTCOMES:
Pathological response | after 13 weeks.
R0 or R1 resection | after 13 weeks.
Postoperative complications (within 8 weeks after surgery) | within 8 weeks after surgery
Time to local relapse | calculated from randomization to documented relapse or censored at the last CT and/or endorectal ultrasound without local relapse.
Time to distant failure | calculated from randomization to documented distant (metastatic) failure or censored at the last CT without distant (metastatic) failure.
Disease-free survival | calculated from randomization to first relapse or death (whichever occurs first).
Adverse events | All AEs will be assessed according to NCI CTCAE v3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Helbling, MD, Study Chair — Onkozentrum Zürich
Locations (24):
- Szent Laszlo Korhaz, Budapest, Hungary
- Switzerland (23):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - OnkoZentrum Luzern at Klinik St. Anna, Lucerne
  - Kantonsspital, Luzerne, Luzerne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital Regional de Sion-Herens-Conthey, Sion
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum, Zurich
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Helbling D, Bodoky G, Gautschi O, Sun H, Bosman F, Gloor B, Burkhard R, Winterhalder R, Madlung A, Rauch D, Saletti P, Widmer L, Borner M, Baertschi D, Yan P, Benhattar J, Leibundgut EO, Bougel S, Koeberle D. Neoadjuvant chemoradiotherapy with or without panitumumab in patients with wild-type KRAS, locally advanced rectal cancer (LARC): a randomized, multicenter, phase II trial SAKK 41/07. Ann Oncol. 2013 Mar;24(3):718-25. doi: 10.1093/annonc/mds519. Epub 2012 Nov 8. PMID 23139259